CLINICAL TRIAL: NCT00285168
Title: A Randomized Controlled Trial of a Bone Density Decision Aide in the Pharmacological Management of Osteoporosis
Brief Title: A Randomized Controlled Trial of a Bone Density Decision Aide
Status: Terminated | Type: Observational
Why Stopped: Inadequate recruitment
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, William D. Leslie, Professor of Medicine and Radiology, University of Manitoba
Other Study IDs: H2003:099
Record Dates: First submitted 2006-01-30; First posted 2006-02-01 (Estimated); Last update posted 2012-07-20 (Estimated); Status verified 2012-07

CONDITIONS: Osteoporosis
Keywords: Osteoporosis; Fractures, Bone; Bone Mineral Density
MeSH Terms: conditions — Osteoporosis; Fractures, Bone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- 1 - Control: Usual Bone Density Report
- 2 - Intervention: Bone Density Report with Absolute 10-year Fracture Risk Decision Aide
  Interventions: Behavioral: Bone Density Decision Aide

INTERVENTIONS:
Behavioral: Bone Density Decision Aide — Absolute 10-year Fracture Risk Report
  Groups: 2 - Intervention

SUMMARY:
This research study is being conducted to determine if a modified bone mineral density (BMD) test report that contains additional fracture risk information will be a useful physician decision aide in selecting patients for pharmacological osteoporosis therapy. It is hypothesized that this supplementary information, provided in addition to the conventional BMD report, will increase the likelihood that patients at high risk for an osteoporotic fracture will receive prescribed therapy for osteoporosis.

DETAILED DESCRIPTION:
This observational research study is being conducted to determine if a modified bone mineral density (BMD) test report that contains additional fracture risk information will be a useful physician decision aide in selecting patients for pharmacological osteoporosis therapy. It is hypothesized that this supplementary information, provided in addition to the conventional BMD report, will increase the likelihood that patients at high risk for an osteoporotic fracture will receive prescribed therapy for osteoporosis. Physicians who only receive the conventional BMD reports without the supplemental information will be the control group.

To compare the rates of pharmacological interventions for osteoporosis in post-menopausal women, family / primary care physicians are randomized to receive either:(i) a conventional BMD report (absolute bone density, T-score result, Z-score result, qualitative statement indicating the BMD results classification of risk for fracture from osteoporosis according to the World Health Organization (WHO) criteria) versus (ii) a conventional BMD report plus a supplemental information sheet (all the information contained in the conventional BMD report plus five-year estimated risks for future fractures calculated from the physician-supplied clinical risk factors and - for those who have osteoporosis according to the WHO criteria - the number needed to treat (in person years) to prevent one fracture.

ELIGIBILITY:
Inclusion Criteria:

* physicians involved in referring patients for DXA bone density testing

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients of physicians involved in referring patients for DXA bone density testing
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2005-05; Primary Completion 2008-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William D Leslie, MD FRCPC, Principal Investigator — University of Manitoba
Locations (1):
- St. Boniface General Hospital, Winnipeg, Manitoba, Canada

REFERENCES:
- See also: Province of Manitoba BMD Program — http://www.gov.mb.ca/health/bonedensity/index.html